CLINICAL TRIAL: NCT00394160
Title: A Randomized, 3-Period, Multiple-Dose, Multicenter Study to Evaluate the Safety, Tolerability, and Plasma Concentration Profile of Montelukast Administered Once Daily as Oral Granules in Children Aged 1 to 3 Months
Brief Title: Safety and Pk Study in 1- to 3- Month-Old Children With Bronchiolitis (0476-297)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-297; 2006_544
Record Dates: First submitted 2006-10-27; First posted 2006-10-31 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-01

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis | interventions — montelukast; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0476, Montelukast Sodium /Duration of Treatment : 14 Days

SUMMARY:
The purpose of this study is to look at the preliminary safety profile of an investigational drug in children 1 to < 3 months of age with bronchiolitis.

ELIGIBILITY:
Inclusion Criteria :

* Active bronchiolitis and a history of bronchiolitis and asthma-like symptoms.

Exclusion Criteria :

* Anemia or history of any significant illness that will pose additional risk to the patient.

Ages: 1 Month to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2004-12; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of montelukast oral granules in children aged 1 to 3 months.

SECONDARY OUTCOMES:
To estimate the single-dose population pharmacokinetics, (maximum plasma concentration, time to maximum plasma concentration, and apparent half-life) of montelukast 4-mg oral granules in children aged 1 to 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Kearns GL, Lu S, Maganti L, Li XS, Migoya E, Ahmed T, Knorr B, Reiss TF. Pharmacokinetics and safety of montelukast oral granules in children 1 to 3 months of age with bronchiolitis. J Clin Pharmacol. 2008 Apr;48(4):502-11. doi: 10.1177/0091270008314251. Epub 2008 Feb 22. PMID 18296556